CLINICAL TRIAL: NCT04681014
Title: Evidence-based Detection of CTEPH in Patients With Prior Pulmonary Embolism: Risk Score Evaluation and Validation.
Brief Title: CTEPH in Patients With Prior Pulmonary Embolism and Risk Score Validation
Acronym: CTEPH-SOLUTION
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: iPHNET (italian Pulmonary Hypertension NETwork) (Other)
Responsible Party: Sponsor
Other Study IDs: CTEPH-SOLUTION
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CTEPH-SOLUTION aims to create a risk score for the early detection of Chronic Thrombo-Embolic Pulmonary Hypertension (CTEPH) among patients with previous pulmonary embolism.

The risk score, created on retrospective data, will be validated on newly diagnosed pulmonary embolism patients.

DETAILED DESCRIPTION:
CTEPH-SOLUTION is a multicenter observational cross-sectional and prospective study in patients with a prior and new diagnosis of pulmonary embolism.

Patients with prior pulmonary embolism will be screened at baseline with doppler echocardiography: an estimated sPAP ≥ 40 mmHg will be the indication for pulmonary hypertension detection. After 24 months from baseline, patients will be followed-up for CTEPH detection. CTEPH diagnosis will be carried out according to the current ESC/ERS guidelines.

Incident (pulmonary embolism episode at least three months before the baseline) and prevalent (pulmonary embolism episode) patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 at baseline evaluation
* Diagnosis of prior (> 30 days from pulmonary embolism onset) or new-onset pulmonary embolism, according to the ESC guidelines on the diagnosis and management of acute pulmonary embolism

Exclusion Criteria:

* patients without pulmonary embolism diagnosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prior pulmonary embolism followed by centres for anticoagulant therapy management (TAO centres) will be enrolled by the investigator's centres and undergo baseline evaluation for prevalent CTEPH detection; al CTEPH will be confirmed by right heart catheterization.
Sampling Method: Probability Sample
Enrollment: 1218 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
CTEPH-SOLUTION score | 24 months
  The CTEPH-SOLUTION score will be created on retrospective parameters (i.e., demographic data, diagnostic and clinical information, risk factors, laboratories parameters) collected on pulmonary embolism patients.
  The minimum and maximum values will be defined after the multivariate statistical analysis, and the risk factors analyzed a posteriori. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The number of the subject with a diagnosis of CTEPH on the total number of subjects enrolled. | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical, Internal, Anesthesiological and Cardiovascular Sciences. AOU Policlinico Umberto I, Rome, Italy